CLINICAL TRIAL: NCT06980493
Title: Efficacy and Safety of Topical Amphotericin B Solution in Treatment of Resistant Tinea Capitis
Brief Title: Efficacy and Safety of Topical Amphotericin B Solution in Treatment of Resistant Tinea Capitis in Children 16 Years Old or Less we Follow up Cases Weekly up to 8 Weeks and Notice Improvement of Itching ,Scaling, and Hair Regrowth Then Fungal Culture Done to See if the Solution Working
Acronym: prospective
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zainab Alkassem Nour, Principal Investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-1-04MS
Record Dates: First submitted 2025-04-28; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Tinea Capitis
Keywords: topical amphotericin b solution in tinea capitis
MeSH Terms: conditions — Tinea Capitis | interventions — Liposomes; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- amphotericin b topical solution (Active Comparator): evaluate the efficacy and safety of topical amphotericin B solution in treatment of non-inflammatory type of tinea capitis after resistant response to oral systemic treatment .
  Interventions: Drug: Amphotericine in liposome (Ambisome®)

INTERVENTIONS:
Drug: Amphotericine in liposome (Ambisome®) — The aim of the study will be to evaluate the efficacy and safety of topical amphotericin B solution in treatment of non-inflammatory type of tinea capitis after resistant response to oral systemic treatment

SUMMARY:
The goal of this clinical trial is to learn if topical amphotericin b solution works to treat resistant cases of tinea capitis in children. It will also learn about the safety of drug. The main questions it aims to answer are:

Does amphotericin b solution effective in cases not cured by systemic antifungal tab?

Participants will:

use topical amphotericin b solution every day for8 weeks Visit the clinic once every 1 week for follow up then follow up after 1 month and fungal culture will be done to test if the treatment working

DETAILED DESCRIPTION:
The aim of the study will be to evaluate the efficacy and safety of topical amphotericin B solution in treatment of non-inflammatory type of tinea capitis after resistant response to oral systemic treatment .

Patient and method After approval of the study by Research and Ethical committee at Sohag faculty of medicine, this study will include group of patients attending the outpatient clinic of Dermatology, venereology and andrology department in Sohag university hospital.

An informed written consent will be obtained from parents of all participants after full explanation of the procedure.

Inclusion criteria:

Children aged < 16 years affected by tinea capitis non inflammatory type who are clinically and dermoscopically confirmed after resistant response to oral systemic treatment for 8 weeks.

Study design : prospective clinical study. Sample Size : 30 participants.

Exclusion criteria:

Patients with inflammatory tinea capitis, kerion or favus. Patients with known hypersensitivity to amphotericin B, other systemic conditions or ongoing use of conflicting medications.

method All recruited children will be submitted to clinical assessment as follows

* Personal history: name, age, sex, residence.
* Family history of similar condition.
* Medical history: received systemic antifungal treatment type, dose and for how long.
* Laporatory investigation :CBC and liver function test.
* Complete general examination. To exclude any systemic diseases.
* Dermatological examination:

Clinical examination:

Description of the lesion (site, size, shape, presence of scales, loss of hair or Lymphadenopathy).

Dermoscopic examination:

Dermoscopic features of tinea capitis non inflammatory type includes

* Comma hairs (short hairs that bend and grow back toward the scalp,resembling a comma)
* Corkscrew hairs (short hairs that are coiled up like a corkscrew)
* Zigzag hairs (short hairs with several bends in them like a zigzag pattern)
* Morse code-like .
* Bent hairs.
* Scales, follicular keratosis, and crusts -Erythema -Broken hairs -Black dots.

Procedure:

Preparation Prepare a 2.5% amphotericin B solution by reconstitute liposomal amphotericin B 50 mg vial in 20 ml distilled water result in a final concentration of 2.5 mg/ml. The resulting solution will be stored in bottles with a dropper and protected from light with aluminum foil.

Application Patients apply the solution to each affected area and briefly let the solution evaporate.

Frequency: Apply once daily. Duration: Continue treatment for 8 weeks or until clinical resolution with dermoscopic confirmation.

Treatment Protocol Baseline assessment. Perform a thorough clinical assessment. Instruct patients/guardians on proper application techniques. Schedule weekly follow-ups for 8 weeks. Monitoring

* Monitor for clinical signs of improvement: reduction in itching, scaling and hair regrowth Weekly for 8 weeks then follow up after 1 month with dermoscopic photographing .
* A fungal culture test will be done in follow up visit after 1 month to test if the treatment is working.
* follow up monitor for side effects: local irritation, redness or systemic reactions

ELIGIBILITY:
Inclusion Criteria:

* Children aged < 16 years affected by tinea capitis non inflammatory type who are clinically and dermoscopically confirmed after resistant response to oral systemic treatment for 8 weeks.

Exclusion Criteria:

* Patients with inflammatory tinea capitis, kerion or favus. Patients with known hypersensitivity to amphotericin B, other systemic conditions or ongoing use of conflicting medications.

Ages: 0 Days to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
monitoring for reduction in size of scaling weekly for 8 weeks | 4 months
  • children 16 years old or less will be evaluated to detect an effect size of 0.3 in the rate of the disease improvement (reduction in scaling) on repeated measurements (follow up weekly for 8 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
result of the study
Supporting Information: Study Protocol